CLINICAL TRIAL: NCT06325124
Title: Effect Of Muscle Energy Technique Of Lower Limb Superficial Backline Muscles in Patients With Forward Head Posture
Brief Title: Muscle Energy Technique of Lower Limb Muscles in Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01805 MARIA NAWAZ
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Forward Head Posture
Keywords: Muscle energy technique; Conventional physical therapy; Superficial backline MUSCLES

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique of Calf and hamstrings (Active Comparator): Muscle Energy Technique of Calf and hamstrings (soft tissue technique)
  Interventions: Other: Muscle energy technique
- Conventional PT (Other): Cervical isometric exercises Hot pack
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Muscle energy technique — They would be receiving treatment as follow:
  Muscle energy technique of hamstring and gastro-soleus. Frequency: 10 reps 3 times/week for 4 consecutive weeks Intensity starting from 20% to 50% resistance across barrier provided by Physical therapist Conventional PT including 1-cervical isometric exercises 2-Transcutaneous Electrical Nerve Stimulation (TENS) for 1o minutes 3-hot pack for 10 minutes 4-Stretching exercise for suboccipitals, sternocleidomastoid 5-gentle stretching of calf and hamstrings.
  Arms: Muscle Energy Technique of Calf and hamstrings
Other: Conventional PT — They would be receiving treatment as follow:
  Conventional PT including 1-cervical isometric exercises 2-Transcutaneous Electrical Nerve Stimulation (TENS) for 1o minutes 3-hot pack for 10 minutes 4-Stretching exercise for suboccipitals, sternocleidomastoid 5-gentle stretching of calf and hamstrings.
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to find the effect of muscle energy technique of muscles involved in lower limb superficial backline (hamstring and Gastro-soleus) on improving craniovertebral angle and cervical proprioception and minimizing pain among patients with forward head posture

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common postural disorder (66%), occurring when the head is anterior to a vertical line passing through the center of gravity. This malalignment causes muscle weakness in deep cervical flexors and shortened opposing cervical extensor muscles. This posture increases lordosis in the lower cervical spine, leading to increased extension over upper, and flexion over the lower cervical spine. Abnormal postures can lead to headaches, myofascial pain syndrome, abnormal scapular movement, temporomandibular disorders, and limited cervical range of motion.

Muscles of the neck, back and lower limb are interconnected through myofascial called superficial backline. Prolonged forward head posture affects muscles and involved in superficial backline. So remote muscle stretching has a same effect on local neck muscles.

Muscle energy technique is a soft tissue technique designed to improve musculoskeletal function through stretching tight muscles and fascia, to reduce pain and improve circulation. MET is characterized by a patient-induced skeletal muscle contraction against physiotherapist resistance in a controlled direction and position. Pathological barrier of a muscle is located through joint positioning which is followed by active muscle contraction by the patient moving away from the resistance followed by relaxation of the muscle. A new pathological barrier is located through passive movement and process is repeated. The rationale for the use of these techniques is to identify the effects of MET of lower limb superficial backline muscles which are interconnected with cervical muscles through myofacial chain, on cervical pain ROM, craniovertebral angle , disability and cervical proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years
* Both Genders
* Craniovertebral angle <49.9 degrees
* History of neck pain >3 months
* Patients with hamstring tightness(Inability to achieve greater than 160° of knee extension with hip at 90° of flexion)
* Patients with calf muscle tightness(The Taloche Sign (Maestro) If a patient with a tight gastrocnemius tries to stand on an inclined plane, it is immediately evident that it is impossible for the patient to be stable in this position)

Exclusion Criteria:

* Patient with recent injuries or surgeries in and around the neck region
* Vertigo
* radiating pain in upper limb
* spinal deformities
* malignancy in and around the neck region
* cervical instabilities
* fibromyalgia
* patients with any lower limb or lower back pathology(e.g arthritis)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Neck disability index (NDI) | 4 weeks
  The NDI is a Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  The NDI is composed of 10 items. Each item consists of different statements which describe how much neck pain interferes with certain activity. Patient choses one option which describes his pain most precisely.
Numeric Pain Rating Scale NPRS | 4 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.

SECONDARY OUTCOMES:
Bubble inclinometer | 4 weeks
  It is an instrument that measures the available range of motion at a joint.
FHP Mobile Application (To measure Craniovertebral angle) | 4 weeks
  FHP app is a free mobile application that enables measurement of the CV angle for the analysis of cervical posture in the sagittal plane. It was used to measure the CV angle. The protocol involved:(1) Preparation of the location of the camera and the subject; (2) palpation and marking anatomical reference points(3) realization of the photographs.
Cervical Joint Position Error | 4 weeks
  The patient is sitting 90 cm from the wall, and the starting point (center of target or reference point) of the laser projection is marked. The patient (blindfolded or closed) performs active neck movement and then returns to the starting position as accurately as possible. The final laser position is measured relative to the starting position (distance or angle). The errors are measured after cervical extension and flexion.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- We Care Physical Therapy Clinic street 13 phase 4A, Ghouri town Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No